CLINICAL TRIAL: NCT03346057
Title: A Phase 4 Randomized, Active-Comparator Controlled Clinical Trial to Study the Safety of Sugammadex (MK-8616) for the Reversal of Neuromuscular Blockade Induced by Either Rocuronium Bromide or Vecuronium Bromide in American Society of Anesthesiologists (ASA) Class 3 or 4 Subjects
Brief Title: Safety of Sugammadex for the Reversal of Neuromuscular Blockade in American Society of Anesthesiologists (ASA) Class 3 or 4 Participants (MK-8616-145)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8616-145; 2017-000187-15 (EudraCT Number); MK-8616-145 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Reversal of Neuromuscular Blockade
Keywords: arrhythmia, bradycardia, neuromuscular blocking agents, surgery, tachycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Tachycardia | interventions — Sugammadex; Neostigmine; Glycopyrrolate; Rocuronium; Vecuronium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sugammadex 2 mg/kg (Experimental): Sugammadex 2 mg/kg administered as a single intravenous (IV) dose
  Interventions: Drug: Sugammadex 2 mg/kg; Drug: Rocuronium; Drug: Vecuronium
- Sugammadex 4 mg/kg (Experimental): Sugammadex 4 mg/kg administered as a single IV dose
  Interventions: Drug: Sugammadex 4 mg/kg; Drug: Rocuronium; Drug: Vecuronium
- Sugammadex 16 mg/kg (Experimental): Sugammadex 16 mg/kg administered as a single IV dose
  Interventions: Drug: Sugammadex 16 mg/kg; Drug: Rocuronium
- Neostigmine + Glycopyrrolate (Active Comparator): Neostigmine 50 μg/kg (up to 5 mg maximum dose) plus glycopyrrolate 10 μg/kg (up to 1 mg maximum dose) administered as a single IV dose
  Interventions: Drug: Neostigmine + Glycopyrrolate; Drug: Rocuronium; Drug: Vecuronium

INTERVENTIONS:
Drug: Sugammadex 2 mg/kg — Following administration of NMBA (Rocuronium or Vecuronium) to achieve moderate NMB, participants received a single i.v. bolus of Sugammadex 2 mg/kg for reversal of moderate NMB. Moderate block is a level of NMB in which peripheral nerve stimulation elicits one to four muscle twitches.
  Other Names: MK-8616; Bridion
  Arms: Sugammadex 2 mg/kg
Drug: Sugammadex 4 mg/kg — Following administration of NMBA (Rocuronium or Vecuronium) to achieve deep NMB, participants received a single i.v. bolus of Sugammadex 4 mg/kg for reversal of deep NMB. Deep block is a level of NMB in which peripheral nerve stimulation elicits no muscle twitches and high-frequency muscle stimulation elicits minimal levels of muscle contraction.
  Other Names: MK-8616; Bridion
  Arms: Sugammadex 4 mg/kg
Drug: Sugammadex 16 mg/kg — Following administration of NMBA (Rocuronium) to achieve deep NMB, participants received a single i.v. bolus of Sugammadex 16 mg/kg for reversal of deep NMB. Deep block is a level of NMB in which peripheral nerve stimulation elicits no muscle twitches and high-frequency muscle stimulation elicits minimal levels of muscle contraction.
  Other Names: MK-8616; Bridion
  Arms: Sugammadex 16 mg/kg
Drug: Neostigmine + Glycopyrrolate — Following administration of NMBA (Rocuronium or Vecuronium) to achieve moderate NMB, participants received a single i.v. bolus of Neostigmine (50 μg/kg; 5 mg maximum) and Glycopyrrolate (10 μg/kg; 1 mg maximum) for reversal of moderate NMB. Moderate block is a level of NMB in which peripheral nerve stimulation elicits one to four muscle twitches.
  Arms: Neostigmine + Glycopyrrolate
Drug: Rocuronium — To achieve NMB, participants received steroidal NMBA Rocuronium Bromide administered via IV infusion and dosed according to participant body weight. NMBAs were concomitant medications used per label and at Investigator's discretion as an adjunct to general anesthesia.
Drug: Vecuronium — To achieve NMB, participants received steroidal NMBA Vecuronium Bromide administered via IV infusion and dosed according to participant body weight. NMBAs were concomitant medications used per label and at Investigator's discretion as an adjunct to general anesthesia.
  Arms: Neostigmine + Glycopyrrolate; Sugammadex 2 mg/kg; Sugammadex 4 mg/kg

SUMMARY:
The purpose of this trial is to evaluate the safety of sugammadex for the reversal of neuromuscular blockade (NMB) induced by neuromuscular blockade agents (NMBA) rocuronium or vecuronium in adult American Society of Anesthesiologists (ASA) Physical Status Class 3 and 4 participants. The primary objectives of the study are to characterize the incidence of treatment emergent sinus bradycardia, treatment emergent sinus tachycardia, or other treatment emergent cardiac arrhythmias after administration of sugammadex and to evaluate the general safety of sugammadex in a population of ASA Class 3 and 4 participants in a surgical setting.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) < 40 kg/m2.
* Is categorized as ASA Physical Status Class 3 or 4, as determined by the Investigator.
* Has a planned surgical procedure that requires NMB with either rocuronium or vecuronium.
* Has a planned surgical procedure (e.g., gastrointestinal, urologic, or laparoscopic) that in the opinion of the investigator does not preclude maintenance of moderate or deep depth of NMB throughout the case.
* If female who is not of reproductive potential, is one of the following: (1) postmenopausal; (2) has had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; (3) has a congenital or acquired condition that prevents childbearing; or (4) is undergoing surgical sterilization (e.g., hysterectomy or tubal ligation) as the planned surgical procedure associated with participation in this study.
* If female who is sexually active and of child-bearing potential, agrees to use a medically accepted method of contraception through seven days after receiving protocol-specified medication. Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and Ethics Review Committees/Institutional Review Boards.
* Is able to provide (or the participant's legally authorized representative, in accordance with local requirements), written informed consent for the trial. The participant or legally authorized representative may also provide consent for Future Biomedical Research.

Exclusion Criteria:

* Has a pacemaker or automatic implantable cardioverter-defibrillator that precludes the assessment of bradycardia or arrhythmias.
* Has a medical condition or surgical procedure that precludes reversal of neuromuscular block at the end of surgery.
* Has a neuromuscular disorder(s) that may affect neuromuscular block and/or trial assessments.
* Is dialysis-dependent or has severe renal insufficiency, defined as estimated creatinine clearance of <30 mL/min.
* Has or is suspected of having a personal history or family history (parents, grandparents, or siblings) of malignant hyperthermia.
* Has or is suspected of having an allergy (e.g., hypersensitivity and/or anaphylactic reaction) to study treatments or its/their excipients, to opioids/opiates, muscle relaxants or their excipients, or other medication(s) used during general anesthesia.
* Has received or is planned to receive toremifene within 24 hours before or within 24 hours after study medication administration.
* Has any condition that would contraindicate the administration of study medication.
* Is pregnant, is attempting to become pregnant, or is lactating.
* Is currently participating in or has participated in an interventional clinical trial (including any other current or ongoing trial with a sugammadex treatment arm) with an investigational compound or device within 30 days of signing the informed consent form of this current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- United States (20):
  - University of Alabama - Birmingham ( Site 1046), Birmingham, Alabama
  - University Banner Medical Center ( Site 1019), Tucson, Arizona
  - Loma Linda University Medical Center ( Site 1029), Loma Linda, California
  - University of California Davis Medical Center ( Site 1001), Sacramento, California
  - Jackson Memorial Hospital ( Site 1007), Miami, Florida
  - University of Kansas Medical Center ( Site 1050), Kansas City, Kansas
  - Tulane University ( Site 1057), New Orleans, Louisiana
  - Ochsner Clinic Foundation ( Site 1005), New Orleans, Louisiana
  - Brigham & Women's Hospital ( Site 1039), Boston, Massachusetts
  - Beaumont Hospital, Royal Oak ( Site 1034), Royal Oak, Michigan
  - University Hospital- Columbia MO ( Site 1060), Columbia, Missouri
  - University of Missouri Health Care ( Site 1022), Columbia, Missouri
  - Jersey Shore University Medical Center ( Site 1058), Neptune City, New Jersey
  - Saint Peter's University Hospital [New Brunswick, NJ] ( Site 1017), New Brunswick, New Jersey
  - Mission Hospital - Memorial ( Site 1016), Asheville, North Carolina
  - Cleveland Clin Foundation ( Site 1032), Cleveland, Ohio
  - Temple University Hospital ( Site 1004), Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center ( Site 1033), Nashville, Tennessee
  - Hermann Drive Surgical Center ( Site 1021), Houston, Texas
  - Zablocki VA Medical Center ( Site 1011), Milwaukee, Wisconsin
- Austria (3):
  - A.O. Krankenhaus Dornbirn ( Site 1151), Dornbirn, Voralberg
  - Landeskrankenhaus Feldkirch ( Site 1152), Feldkirch
  - Sozialmedizinisches Zentrum Ost - Donauspital ( Site 1150), Vienna
- Denmark (4):
  - Aarhus Universitets hospital ( Site 1252), Aarhus
  - Rigshospitalet ( Site 1253), Copenhagen
  - Bispebjerg og Frederiksberg Hospital ( Site 1250), Copenhagen NV
  - Regionshospitalet Viborg ( Site 1254), Viborg
- Germany (3):
  - Klinikum Rechts der Isar Technische Universitaet Muenchen ( Site 1350), München
  - Klinikum am Steinenberg Reutlingen ( Site 1352), Reutlingen
  - Josephs-Hospitals Warendorf ( Site 1351), Warendorf

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Herring WJ, Mukai Y, Wang A, Lutkiewicz J, Lombard JF, Lin L, Watkins M, Broussard DM, Blobner M. A randomized trial evaluating the safety profile of sugammadex in high surgical risk ASA physical class 3 or 4 participants. BMC Anesthesiol. 2021 Oct 28;21(1):259. doi: 10.1186/s12871-021-01477-5. PMID 34711192

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 344 participants randomized to the study, 331 received at least one dose of study treatment (All Treated Population) and were evaluable for all safety analysis.
Period: Overall Study
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Started | 111 | 112 | 68 | 53
Treated | 105 | 107 | 68 | 51
Completed | 104 | 104 | 67 | 51
Not Completed | 7 | 8 | 1 | 2
Not completed — Death | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0
Not completed — Ineligible For Study - Not Treated | 0 | 1 | 0 | 0
Not completed — Renal Insufficiency - Not Treated | 1 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 0 | 2
Not completed — Randomization Mistake - Not Treated | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate | Total
Number analyzed (Participants) | 111 | 112 | 68 | 53 | 344
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.5 (10.7) | 67.8 (12.1) | 69.4 (10.0) | 66.6 (10.9) | 68.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 41 | 29 | 15 | 135
  Male | 61 | 71 | 39 | 38 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 0 | 2 | 10
  Not Hispanic or Latino | 109 | 105 | 67 | 51 | 332
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 3 | 9 | 2 | 3 | 17
  White | 106 | 103 | 66 | 50 | 325
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Participant Stratifications [Count of Participants; unit: Participants] — Participants were stratified by neuromuscular blockade agent (NMBA, rocuronium or vecuronium) and American Society of Anesthesiologists (ASA) Class which ranges from ASA 1 (Normal healthy patient) to ASA 6 (Declared brain-dead patient whose organs are being removed for donor purposes). Higher ASA class with other factors (surgery type, frailty, and deconditioning) help predict greater perioperative risk. Participants were graded as ASA 3 if participants had severe systematic disease and as ASA 4 if participants had severe systematic disease that was a constant threat to the life.
  Participants
    Rocuronium, ASA Class 3 | 50 | 49 | 51 | 25 | 175
    Rocuronium, ASA Class 4 | 15 | 18 | 17 | 8 | 58
    Vecuronium, ASA Class 3 | 29 | 31 | 0 | 14 | 74
    Vecuronium, ASA Class 4 | 11 | 11 | 0 | 5 | 27
    Missing | 6 | 3 | 0 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Sinus Bradycardia Events
Description: The percentage of participants experiencing treatment-emergent sinus bradycardia events was identified with continuous electrocardiogram (ECG) monitoring. Treatment-emergent sinus bradycardia were defined as a heart rate <60 bpm that has also decreased more than 20% compared to participant baseline heart rate value, sustained for at least 1 minute after administration of study intervention. Treatment-emergent sinus bradycardia events may or may not have been considered an adverse event (AE), as determined by investigator judgment.
Time Frame: Up to approximately 35 minutes post-administration
Population: All randomized participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Number analyzed (Participants) | 105 | 107 | 68 | 51
Percentage of participants | 1.0 | 1.9 | 7.4 | 7.8
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg vs Neostigmine + Glycopyrrolate; Miettinen & Nurminen method stratified by neuromuscular blocking agent (NMBA) and American Society of Anesthesiologists (ASA) class was used to provide estimated between-treatment difference, 95% confidence interval, and p-value; Test type: Other; p = 0.026, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -6.7, 95% CI 2-sided [-17.5 to -0.8]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Neostigmine + Glycopyrrolate; Miettinen & Nurminen method stratified by NMBA and ASA was used to provide estimated between-treatment difference, 95% confidence interval, and p-value; Test type: Other; p = 0.058, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -6.2, 95% CI 2-sided [-17.3 to 0.2]
Statistical Analysis 3: Comparison: Sugammadex 16 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.730, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -2.0, 95% CI 2-sided [-17.8 to 8.6]

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Sinus Tachycardia Events
Description: The percentage of participants experiencing treatment-emergent sinus tachycardia events was identified with continuous ECG monitoring. Treatment-emergent sinus tachycardia is defined as a heart rate ≥100 bpm that has also increased more than 20% compared to participant baseline heart rate value, sustained for at least 1 minute after administration of study intervention. Treatment-emergent sinus tachycardia events may or may not have been considered an AE, as determined by investigator judgment.
Time Frame: Up to approximately 35 minutes post-administration
Population: All randomized participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Number analyzed (Participants) | 105 | 107 | 68 | 51
Percentage of participants | 6.7 | 9.3 | 8.8 | 21.6
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.007, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -14.9, 95% CI 2-sided [-28.8 to -4.0]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.036, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -12.2, 95% CI 2-sided [-26.1 to -0.8]
Statistical Analysis 3: Comparison: Sugammadex 16 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.158, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -9.9, 95% CI 2-sided [-27.6 to 3.6]

3. Primary Outcome: Percentage of Participants With Other Treatment-Emergent Cardiac Arrhythmia Events
Description: The percentage of participants experiencing other treatment-emergent cardiac arrhythmia events was identified with continuous ECG monitoring. Other treatment-emergent cardiac arrhythmias were defined as new or worsening arrhythmias (e.g., atrial fibrillation, atrial tachycardia, ventricular fibrillation, or ventricular tachyarrhythmia), sustained for at least 1 minute after administration of study intervention. Worsening arrhythmia events may or may not have been considered an AE, as determined by investigator judgment.
Time Frame: Up to approximately 35 minutes post-administration
Population: All randomized participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Number analyzed (Participants) | 105 | 107 | 68 | 51
Percentage of participants | 1.0 | 0.0 | 1.5 | 2.0
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.637, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -0.9, 95% CI 2-sided [-9.4 to 4.0]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.134, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -2.1, 95% CI 2-sided [-10.6 to 1.5]
Statistical Analysis 3: Comparison: Sugammadex 16 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.577, Stratified Miettinen & Nurminen method; Estimated Difference in percentage = -1.7, 95% CI 2-sided [-14.7 to 5.8]

4. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE) Up To 7 Days After Administration of Study Intervention
Description: As per the protocol primary analysis, the percentage of participants experiencing an AE up to 7 days after administration of study intervention was reported. An AE was defined as any untoward medical occurrence in a participant which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE.
Time Frame: Up to 7 days
Population: All randomized participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Number analyzed (Participants) | 105 | 107 | 68 | 51
Percentage of participants | 94.3 | 88.8 | 92.6 | 88.2
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg vs Neostigmine + Glycopyrrolate; Miettinen & Nurminen method stratified by NMBA and ASA was used to provide estimated between-treatment difference and 95% confidence interval; Test type: Other; Estimated Difference in percentage = 6.2, 95% CI 2-sided [-2.6 to 18.5]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 4, analysis 1]; Test type: Other; Estimated Difference in percentage = 0.5, 95% CI 2-sided [-9.3 to 13.1]
Statistical Analysis 3: Comparison: Sugammadex 16 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 4, analysis 1]; Test type: Other; Estimated Difference in percentage = 2.0, 95% CI 2-sided [-8.4 to 17.7]

5. Primary Outcome: Percentage of Participants Experiencing a Serious Adverse Event (SAE) Up To 7 Days After Administration of Study Intervention
Description: As per the protocol primary analysis, the percentage of participants experiencing an SAE up to 7 days after administration of study intervention was reported. An SAE was an adverse event that: resulted in death; was life threatening; resulted in persistent or significant disability or incapacity; resulted in or prolonged an existing inpatient hospitalization; was a congenital anomaly or birth defect; was an other important medical event, was a cancer; or was associated with an overdose.
Time Frame: Up to 7 days
Population: All randomized participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Number analyzed (Participants) | 105 | 107 | 68 | 51
Percentage of Participants | 11.4 | 7.5 | 10.3 | 5.9
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 4, analysis 1]; Test type: Other; Estimated Difference in percentage = 5.6, 95% CI 2-sided [-5.5 to 14.3]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 4, analysis 1]; Test type: Other; Estimated Difference in percentage = 1.5, 95% CI 2-sided [-9.2 to 9.3]
Statistical Analysis 3: Comparison: Sugammadex 16 mg/kg vs Neostigmine + Glycopyrrolate; [analysis description as in outcome 4, analysis 1]; Test type: Other; Estimated Difference in percentage = 0.9, 95% CI 2-sided [-15.1 to 12.7]

6. Primary Outcome: Percentage of Participants Experiencing an Event of Clinical Interest (ECI) Up To 7 Days After Administration of Study Intervention
Description: As per the protocol primary analysis, the percentage of participants experiencing an ECI up to 7 days after administration of study intervention was reported. ECIs were a discrete set of both AEs and SAEs, specifically designated as such for the trial. For the purposes of this investigation, ECIs included 1) drug-induced liver injury; 2) clinically-relevant arrhythmias, inclusive of bradycardia and tachycardia defined as events necessitating intervention, as determined by investigator judgment; and 3) instances of hypersensitivity and/or anaphylaxis adjudicated by an external expert Adjudication Committee. A participant could have experienced more than one type of ECI.
Time Frame: Up to 7 days
Population: All randomized participants who received at least one dose of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
Number analyzed (Participants) | 105 | 107 | 68 | 51
Percentage of Participants
  With one or more ECIs | 1.9 | 5.6 | 7.4 | 3.9
  Adjudicated Hypersensitivity | 0.0 | 0.0 | 0.0 | 0.0
  Adjudicated Anaphylaxis | 0.0 | 0.0 | 0.0 | 0.0
  Clinically Relevant Bradycardia | 0.0 | 2.8 | 0.0 | 2.0
  Clinically Relevant Tachycardia | 1.9 | 1.9 | 5.9 | 0.0
  Other Clinically Relevant Cardiac Arrhythmia | 0.0 | 0.9 | 1.5 | 2.0
  Drug Induced Liver Injury | 0.0 | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: Sugammadex 2 mg/kg vs Neostigmine + Glycopyrrolate; The percentage of participants experiencing one or more ECIs was compared between the Sugammadex 2 mg/kg arm and the Neostigmine plus Glycopyrrolate arm. Miettinen & Nurminen method stratified by NMBA and ASA was used to provide estimated between-treatment difference and 95% confidence interval; Test type: Other; Estimated Difference in percentage = -2.1, 95% CI 2-sided [-11.8 to 3.8]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Neostigmine + Glycopyrrolate; The percentage of participants experiencing one or more ECIs was compared between the Sugammadex 4 mg/kg arm and the Neostigmine plus Glycopyrrolate arm. Miettinen & Nurminen method stratified by NMBA and ASA was used to provide estimated between-treatment difference and 95% confidence interval; Test type: Other; Estimated Difference in percentage = 1.8, 95% CI 2-sided [-8.1 to 8.4]
Statistical Analysis 3: Comparison: Sugammadex 16 mg/kg vs Neostigmine + Glycopyrrolate; The percentage of participants experiencing one or more ECIs was compared between the Sugammadex 16 mg/kg arm and the Neostigmine plus Glycopyrrolate arm. Miettinen & Nurminen method stratified by NMBA and ASA was used to provide estimated between-treatment difference and 95% confidence interval; Test type: Other; Estimated Difference in percentage = 1.1, 95% CI 2-sided [-13.5 to 11.1]

ADVERSE EVENTS:
Time Frame: Up to approximately 21 days post treatment
Description: All-Cause Mortality reported for all randomized participants (N = 344: Sugammadex 2 mg/kg: n = 111, Sugammadex 4 mg/kg: n = 112, Sugammadex 16 mg/kg: n = 68, and Neostigmine + Glycopyrrolate: n = 53). Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Sugammadex 2 mg/kg | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Neostigmine + Glycopyrrolate
All-Cause Mortality (participants affected / at risk) | 1/111 | 2/112 | 0/68 | 0/53
Serious Adverse Events (participants affected / at risk) | 16/105 | 12/107 | 9/68 | 4/51
Other Adverse Events (participants affected / at risk) | 89/105 | 89/107 | 60/68 | 41/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 2 mg/kg (N=105) | Sugammadex 4 mg/kg (N=107) | Sugammadex 16 mg/kg (N=68) | Neostigmine + Glycopyrrolate (N=51)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehiscence (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purulent discharge (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fascial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 2 mg/kg (N=105) | Sugammadex 4 mg/kg (N=107) | Sugammadex 16 mg/kg (N=68) | Neostigmine + Glycopyrrolate (N=51)
Bradycardia (Cardiac disorders) | 4 (4) | 4 (4) | 1 (1) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (3) | 5 (5) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (5) | 8 (8) | 3 (3) | 4 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (7) | 6 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 17 (18) | 19 (20) | 13 (14) | 7 (8)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (3) | 2 (4)
Asthenia (General disorders) | 2 (2) | 6 (6) | 2 (2) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 25 (26) | 31 (31) | 19 (19) | 9 (9)
Postoperative hypertension (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 5 (5) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 58 (66) | 56 (67) | 31 (38) | 27 (31)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 5 (5) | 2 (2) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 8 (8) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (4) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 6 (8) | 6 (6) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 6 (6) | 8 (8) | 5 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03346057/Prot_SAP_000.pdf